CLINICAL TRIAL: NCT00532428
Title: Long-Term Effects of Raloxifene Treatment on Bone Quality: A Cross-Sectional Study of Postmenopausal Women With Osteoporosis Previously Enrolled in the Continuing Outcomes Relevant to Evista Study
Brief Title: Long Term Effects of Raloxifene Treatment on Bone Quality
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8149; H3S-MC-GGLF
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Osteoporosis, Post-Menopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Raloxifene Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: Raloxifene
- 2 (Active Comparator)
  Interventions: Drug: Raloxifene
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Raloxifene — 60 mg QD
  Other Names: LY139481
  Arms: 1
Drug: Raloxifene — 120 mg QD
  Other Names: LY139481
  Arms: 2
Drug: Placebo — Placebo
  Arms: 3

SUMMARY:
This is a cross-sectional study to determine, via iliac crest bone biopsies, the effect of long-term treatment with raloxifene on histomorphometry and bone quality in patients who participated in the Continuing Outcomes Relevant to Evista Study.

ELIGIBILITY:
Inclusion Criteria:

* Have completed the CORE protocol within 3 months (90 days) prior to study entry and enrollment.
* Have taken randomized study material for at least 7 years since enrollment in the MORE protocol. If the patient opted not to receive randomized study material for a period of 6 months at any point during either the MORE or CORE protocol, this period must have occurred in its entirety before Visit 3 of the CORE protocol.
* Overall, were at least 75% compliant with randomized study material during the MORE and CORE protocols.

Exclusion Criteria:

* Have an allergy or other intolerance to tetracycline hydrochloride that would preclude its administration in conjunction with the bone biopsy procedures. If the patient is not allergic to all tetracyclines, then this exclusion may be waived by the sponsor and a different tetracycline to which the patient is not allergic may be used.
* Have undergone two previous transiliac bone biopsies (one in each iliac crest). Patients with one previous transiliac bone biopsy are eligible provided that the new sample is obtained from the contralateral iliac crest.
* In the opinion of the investigator, have any medical or anatomical condition that potentially could put the patient at additional risk of an adverse event due to the procedure (for example, coagulation abnormality, extreme obesity, etc.).
* Have a history of bone metabolic diseases, Paget's disease, renal osteodystrophy, osteomalacia, any secondary causes of osteoporosis, hyperparathyroidism (uncorrected), and intestinal malabsorption.
* Have a history of malignant neoplasms in the prior 5 years, with the exception of superficial basal cell carcinoma or squamous cell carcinoma of the skin that has been definitively treated. If malignant neoplasm was ever diagnosed, patient must presently be free of disease.

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2003-04; Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
To determine the histomorphometric effects on bone,by iliac crest bone biopsy, of long-term (7 &8 yrs) therapy with raloxifene or placebo in postmenopausal women with osteoporosis who were enrolled in the CORE trial | 6 months

SECONDARY OUTCOMES:
Find effect of long-term treatment with raloxifene or placebo on bone quality. Primary measures: primary mineralization defect absence, mean degree of mineralization of bone tissue, absence of woven bone, microCT, microcrack & nanoindentation analysis. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City, Mexico
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam, Netherlands
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Granada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oviedo

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com